CLINICAL TRIAL: NCT01668914
Title: Phase III Trail of Internal Mammary Sentinel Lymph Node Biopsy in Early Breast Cancer Patients With Clinically Axillary Node -Positive
Brief Title: Internal Mammary Sentinel Lymph Node Biopsy in Early Breast Cancer Patients With Clinically Axillary Node -Positive
Acronym: IMSLNB-CANP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Yongsheng Wang, Director, Head of Breast Cancer Center, Principal Investigator, Clinical Professor, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IMSN002
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Clinically Axillary Node -Positive; Sentinel Lymph Node Biopsy; Internal Mammary
MeSH Terms: conditions — Breast Neoplasms | interventions — Histological Techniques; Immunohistochemistry; Lymphoscintigraphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- clinically positive axillary nodes (Experimental): 3~18 hours before surgery, under ultrasonographic guidance, 0.5~1.0 mCi 99mTc-SC in sterile saline (total volume 0.2~2.0 mL) is injected intraparenchymally into 2 quadrants of breast. Subsequently, LSG is performed 0.5~1.0 hour before surgery. Methylthioninium was injected intraparenchymally. IM-SLNB is performed during the surgery and the IMSLNs were sent to histologic examination
  Interventions: Procedure: IM-SLNB; Radiation: 99mTc-SC; Device: Histologic Examination; Device: LSG; Drug: Methylthioninium

INTERVENTIONS:
Procedure: IM-SLNB — IM-SLNB is performed according to the pre-operative lymphoscintigraphy
  Other Names: Internal Mammary Sentinel Lymph Node Biopsy
Radiation: 99mTc-SC — Two syringes of 0.25~0.5 mCi 99mTc-SC in 0.2~1.0 mL volume were injected intraparenchymally into 2 quadrants of breast, at the 6 and 12 o'clock positions.
  Other Names: 99mTc-labeled Sulfur Colloid
Device: Histologic Examination — All IMSLNs were analyzed by histologic examination for future therapy planning.
  Other Names: hematoxylin-eosin staining and immunohistochemistry
Device: LSG — lymphoscintigraphy was performed 0.5~1.0 hour before surgery
  Other Names: Lymphoscintigraphy
Drug: Methylthioninium — Four milliliters of methylthioninium was injected intraparenchymally around the primary tumor 10 min before surgery

SUMMARY:
In addition to the axillary lymph nodes, the internal mammary lymph nodes (IMLNs) drainage is another important lymphatic channel of the breast. The status of IMLNs also provides important prognostic information for breast cancer patients. The technical evolvements of sentinel lymph node biopsy (SLNB) and lymphoscintigraphy provided a less invasive method for assessing IMLNs than surgical dissection. Recently, many study concerning IMSLNB was performed in the patients with clinically negative axillary nodes. However, previous published studies concerning patients with breast cancer who all underwent a radical mastectomy have shown that IMLN metastases are mostly found concomitantly with axillary metastases. For this reason, IM-SLNB is even more important for clinically axillary node-negative patients. To our knowledge, this is the first attempt of the IM-SLNB in early breast cancer patients with clinically positive axillary nodes.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the impact of routinely performed internal mammary sentinel lymph node biopsy on the systemic and locoregional treatments plan.
* Evaluate the metastasis rate of internal mammary sentinel lymph nodes in patients with clinically axillary node-positive.
* Draw the learning curve of internal mammary sentinel lymph node biopsy.

OUTLINE:

3~18 hours before surgery, under ultrasonographic guidance, 0.5~1.0 mCi 99mTc-labeled sulfur colloid in sterile saline (total volume 0.2~2.0 mL) is injected intraparenchymally into 2 quadrants of breast. Subsequently, lymphoscintigraphy is performed 0.5~1.0 hour before surgery. internal mammary sentinel lymph node biopsy is performed during the surgery and the internal mammary sentinel lymph nodes were sent to histologic examination.

ELIGIBILITY:
Inclusion Criteria:

* primary breast cancer
* clinically axilla-positive

Exclusion Criteria:

* enlarged internal mammary nodes by imaging

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants Whose Lymph Node Staging was Changed with IM-SLNB | 1 year
  Number of Participants Whose Lymph Node Staging was Changed with IM-SLNB

SECONDARY OUTCOMES:
Visualization Rate of IMSLNs | 1 year
  visualization rate of internal mammary hotspots in lymphoscintigraphy
Metastasis Rate of IMSLNs | 1 year
  Metastasis Rate of internal mammary sentinel lymph node

CONTACTS AND LOCATIONS:
Overall Officials: Yong-sheng Wang, MD, Study Chair — Shandong Cancer Hospital and Institute; Peng-fei Qiu, MD, Principal Investigator — Shandong Cancer Hospital and Institute; Yan-bing Liu, MD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital, Jinan, Shandong, China